CLINICAL TRIAL: NCT02115620
Title: Demonstration Project Using Technology to Improve Health Outcomes for Hospitalized Patients With Heart Failure Discharged to Skilled Nursing Homes
Brief Title: Telemedicine Technology Demonstration Project for Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Verizon Wireless (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-165A
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac failure; Congestive Heart Failure; Cardiomyopathy; Myocardial Failure; Telemedicine; Telehealth; Remote Consultation
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemedicine (Experimental): Patients will be followed using frequent communication of symptom status and physiologic data and remote consultations with Heart Failure specialists.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Daily updates on symptoms, weight, vital signs, and relevant labs will be communicated by phone with cardiology nurses at Providence Heart Clinic. Concerning changes in symptoms or signs will trigger a telemedicine clinic visit with a HF specialist using remote video/audio, virtual stethoscope technology, and VZ Cloud managed hosting. The consult will include a virtual face-face interview and physical examination between patient and HF clinician using Cisco Yabber Video, Littman e-stethoscope, and Verizon managed hosting. Medication changes, laboratory testing, additional virtual visits, or in-person clinic visits can be arranged as appropriate.

SUMMARY:
The purpose of this study is to see if telemedicine can help improve the health of patients with heart failure who have recently been hospitalized with heart problems, and are being discharged to a Skilled Nursing Facility. Telemedicine uses electronic communications to make patient/doctor visits possible from a distance.

This study will use remote video to allow heart failure specialists at Providence St. Vincent Medical Center to provide clinical health care to patients at Marquis Hills. Electronic monitors (including an electronic scale and blood pressure machine), and phone calls with the Marquis Hill nursing staff will be used to track patients' health status. The nursing staff will provide the heart failure specialists with daily updates on patients' symptoms, weight, vital signs (heart rate, blood pressure, pulse), and results of blood tests.

Additionally, some patients will be provided with monitoring devices that include an iPhone blood pressure monitor, and Smart Body Analyzer to use for 14 days. The Smart Body Analyzer measures weight, body fat percentage, and heart rate. It also measures indoor air quality. Special software on the iPhone will save this information and the information will be transmitted by secure email to the study doctors.

Hypothesis: The patients followed by telemedicine will have fewer visits to the Emergency Department, fewer deaths, and fewer hospital re-admissions than last year's site-specific average for this patient population.

DETAILED DESCRIPTION:
The clinical course of heart failure (HF) is highly variable, but most patients eventually require hospitalization to manage symptomatic exacerbations. As HF progresses, hospitalizations become increasingly frequent as overall function and health decline. After an acute hospitalization, many older patients are discharged to skilled nursing facilities (SNF). Patients discharged to SNF after a HF hospitalization experience rates of death and re-hospitalization that are substantially higher than similar patients who are discharged home, even after adjusting for patient factors. The risk of worsening HF is highest in the first week after hospital discharge. Close monitoring of a patient during this vulnerable period could allow early detection and treatment that would avert clinical deterioration and the need for re-hospitalization; however, patients do not routinely receive cardiac specialty care while in SNF for many reasons, including patient immobility, limited transportation options, under-trained staff, competing medical conditions, and lack of timely access to cardiologists.

This research will address the issues associated with heart failure using a multi-faceted intervention consisting of provider, patient, and caregiver education and training, peer-to-peer telephone support for SNF staff, improved access to specialty care to include telemedicine evaluation by HF specialists, and early follow-up following SNF discharge. Specifically: Study the effect of a telemedicine disease management intervention in older patients with HF (either as a primary OR secondary diagnosis) discharged to a SNF from Providence St. Vincent Medical Center (PSVMC) after a cardiac-related admission.

Multiple benefits are anticipated from these interventions. First, a close partnership between the staff at the SNF (Marquis Hills) and the Providence Heart Clinic will be fostered. A major focus early in this partnership will be teaching SNF personnel how to assess signs and symptoms of HF, how to promote patient education and self-management ("teaching the teachers"), and how to use an existing HF disease management tool ("HF Zone tool"). Second, heightened monitoring of patients during the period of greatest risk for HF decompensation is expected to improve care, efficiency, and patient outcomes and reduce costs. Earlier detection and intervention can mitigate worsening HF, as well common complications of HF therapies, such as kidney dysfunction and electrolyte abnormalities. Third, this novel use of telemedicine could radically alter the approach to chronic disease management in care facilities, where specialty care is not readily available even for a high-risk population. Fourth, the use of telemedicine enables the intervention to be scaled easily to other SNFs and clinics and other chronic conditions.

Patients being discharged to Marquis Hills SNF will be identified by case management prior to discharge and consented for enrollment in the study. A Heart Failure clinician, will assess the patient's baseline capacity for self-care for HF (Self Care of Heart Failure Index, SCHFI), and quality of life (Kansas City Cardiomyopathy Questionnaire, KCCQ).

Intake and data collection at SNF will involve baseline assessment of HF symptoms and basic physiologic parameters (weight, blood pressure, heart rate) using the HF Zone tool. Certified nursing assistants will provide basic education on management of heart failure to patient and their families. The first business day following SNF admission, cardiology nurses will contact the SNF staff to review the daily HF Zone tool findings and follow-up any laboratory testing.

Daily updates on symptoms, weight, vital signs, and relevant labs will be communicated by phone with cardiology nurses at Providence Heart Clinic. Concerning changes in symptoms or signs will trigger a telemedicine clinic visit with a HF specialist using remote video/audio, virtual stethoscope technology, and VZ Cloud managed hosting. Any significant changes in symptoms (as reflected by Zone tool) or vital signs will be communicated by cardiology nursing staff to a HF clinician.Within 24 hours of this notification, a telemedicine evaluation will be performed, allowing for a virtual face-face interview and physical examination between patient and HF clinician using Cisco Yabber Video, Littman e-stethoscope, and Verizon managed hosting. Medication changes, laboratory testing, additional virtual visits, or in-person clinic visits can be arranged as appropriate. The visit findings will become part of the patient's electronic medical record and communicated to the facility physician and the patient's outpatient primary care provider.

Upon discharge from the SNF, the patient will have an in-person cardiology follow-up clinic visit within two weeks of discharge and as needed, with re-measurement of the SCHFI at the first follow-up visit.

Subjects' participation in the study will last about 60 days after they are discharged from the skilled nursing facility. They will not be told the results of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary diagnosis of heart failure
* Being discharged to a skilled nursing facility

Exclusion Criteria:

* Life expectancy of < 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03-23 (Actual); Primary Completion 2015-08-26 (Actual); Study Completion 2015-08-26 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (re-admission/ Emergency Department visit/ death) | up to 60 days after patient is discharged from skilled nursing facility
  The primary composite outcome of all-cause re-admission to the hospital/ Emergency Department visits/ death at 30 and 60 days will be compared to facility-specific historical event rates from the prior year.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Abraham, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence St. Vincent Medical Center, Portland, Oregon, United States